CLINICAL TRIAL: NCT03639883
Title: A Randomized, Double-blind, Vehicle-controlled, Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Intradermally Administered AIV001 in Healing of Incisional Wounds
Brief Title: A Safety and Efficacy Study to Evaluate AIV001 in Wound Healing Following Surgical Incision
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AiViva BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AIV001-W01
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Scar; Incision; Abdominal; Wound (Morphologic Abnormality)
Keywords: wound healing; Scar; abdominoplasty
MeSH Terms: conditions — Cicatrix; Surgical Wound; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, vehicle-controlled, dose-escalation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treating investigator will administer the study medication. Evaluating Investigator will perform the safety and efficacy evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.033% versus Vehicle (Experimental): One side of the subject will receive 0.033% AIV001 and the other side of the subject will receive vehicle.
  Interventions: Drug: AIV001
- 0.1% versus Vehicle (Experimental): One side of the subject will receive 0.1% AIV001 and the other side of the subject will receive vehicle.
  Interventions: Drug: AIV001
- 0.3% versus Vehicle (Experimental): One side of the subject will receive 0.3% AIV001 and the other side of the subject will receive vehicle.
  Interventions: Drug: AIV001
- 1% versus Vehicle (Experimental): One side of the subject will receive 1% AIV001 and the other side of the subject will receive vehicle.
  Interventions: Drug: AIV001

INTERVENTIONS:
Drug: AIV001 — Intradermal injection
  Other Names: AIV001 suspension

SUMMARY:
To evaluate the safety, efficacy and pharmacokinetic profile of ascending concentrations of the study medication compared with vehicle in subjects with incisional wounds

DETAILED DESCRIPTION:
This is primarily a safety study to evaluate the safety of AIV001 when administered near incisional wounds. A unique model was used to assess incisional scarring, safety and biomarker assessments. Women electing to have the abdominoplasty procedure were enrolled in the study and abdominal incisions were generated on the abdominal skin. Up to 10 incisions were made on abdominal skn and treated as assigned. And data collection was conducted up to day 49 when the subjects were exited from the study and the abdominoplasty procedure performed. Exploratory efficacy measures were collected and pharmacokinetic profiles determined.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for an abdominoplasty
* Nonsmoker
* Fitzpatrick I-IV
* Weight >45Kg
* BMI <= 35

Exclusion Criteria:

* Existing scars in study area, active infection
* Any medical history or present conditions that may increase the risk associated with study participation or investigational product administration and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Adverse events | Day 1 through Day 49
  Local and systemic adverse events

SECONDARY OUTCOMES:
Efficacy using Patient and Observer Scar Assessment Scale (6 parameters, 1 normal to 10 worst imaginable) | Day 7 through 49
  Evaluation of the healing of the wounds
Modified Vancouver Scar Scale (4 parameters, 0 = normal to 3 or 4 = severe) | Day 7 through 49
  Evaluation of the healing wounds
100 mm Visual Analogue Scale (0 = normal to 10 = poor scar) | Day 7 through 49
  Evaluation of healing wounds

CONTACTS AND LOCATIONS:
Overall Officials: James Milbauer, MD, Study Director — Novella Clinical
Locations (2):
- United States (2):
  - Kaufman and Davis Plastic Surgery, Folsom, California
  - Cosmetic Laser Dermatology, San Diego, California

IPD SHARING:
Plan to Share IPD: No